CLINICAL TRIAL: NCT00707967
Title: Safety and Immunogenicity of a Candidate Tuberculosis (TB) Vaccine (692342) in HIV-positive Adults.
Brief Title: Safety and Immunogenicity of a Candidate Tuberculosis (TB) Vaccine in HIV-positive Adults.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 111517
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2016-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group A (Experimental): Subjects receiving the candidate vaccine
  Interventions: Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342
- Group B (Placebo Comparator): Subjects receiving the adjuvant
  Interventions: Biological: Control vaccine with the adjuvant system.
- Group C (Placebo Comparator): Subjects receiving physiological saline
  Interventions: Biological: Control vaccine with physiological saline

INTERVENTIONS:
Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342 — Intramuscular injection, 2 doses at 0, 1 month
  Arms: Group A
Biological: Control vaccine with the adjuvant system. — Intramuscular injection, 2 doses at 0, 1 month
  Arms: Group B
Biological: Control vaccine with physiological saline — Intramuscular injection, 2 doses at 0, 1 month
  Arms: Group C

SUMMARY:
This study will assess the safety and immunogenicity of a GSK Biologicals' candidate TB vaccine (692342) administered at 0, 1 month to HIV-positive adults living in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the Investigator believes that they can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 50 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to any study procedure.
* Subjects must be HIV-positive and must have:

  * received Highly Active Antiretroviral therapy for a minimum of 12 consecutive months prior to screening
  * documented suppressed HIV-1 RNA levels following HAART-treatment.
  * a protocol defined CD4+ T cell count at screening
* If the subject is female, she must be of non-childbearing potential, or she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of vaccination.
* Clinically acceptable laboratory values prior to randomisation as determined by the Investigator.
* No evidence of TB disease with no pulmonary pathology as confirmed by chest X-ray.
* No history of extrapulmonary TB.
* No history of chemotherapy for TB.

Exclusion Criteria:

* Any change in antiretroviral drug regimen within 12 weeks prior to screening.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of a registered live vaccine not foreseen by the study within 30 days preceding the first dose of study vaccine and administration of a registered inactivated vaccine within 14 days preceding the first dose of study vaccine.
* History of previous administration of experimental Mycobacterium tuberculosis vaccines.
* History of previous exposure to experimental products containing components of the experimental vaccine.
* Chronic administration of immunosuppressive or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of any immunoglobulins, any immunotherapy and/or any blood products within the three months preceding the first dose of study vaccination, or planned administrations during the study period.
* Any condition or illness (acute, chronic or history) or medication, which in the opinion of the Investigator might interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Planned participation or participation in another experimental protocol during the study period.
* A family history of congenital or hereditary immunodeficiency. •Any chronic drug therapy, other than HAART or prophylaxis for opportunistic HIV-related infections to be continued during the study period. Vitamins and/or dietary supplements, birth control pills, anti-histamines for seasonal allergies and SSRIs are allowed.
* Subjects taking any of the following medication: systemic steroids, interleukins, systemic interferons or systemic chemotherapy.
* History of allergic reactions or anaphylaxis to any vaccine.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of chronic alcohol consumption and/or drug abuse which in the Investigator's opinion would put the subject at risk.
* Pregnant female, lactating female or female planning to become pregnant or stop contraception.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-06-30; Primary Completion 2009-05-27 (Actual); Study Completion 2009-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lausanne, Switzerland

REFERENCES:
- [Derived] Thacher EG, Cavassini M, Audran R, Thierry AC, Bollaerts A, Cohen J, Demoitie MA, Ejigu D, Mettens P, Moris P, Ofori-Anyinam O, Spertini F. Safety and immunogenicity of the M72/AS01 candidate tuberculosis vaccine in HIV-infected adults on combination antiretroviral therapy: a phase I/II, randomized trial. AIDS. 2014 Jul 31;28(12):1769-81. doi: 10.1097/QAD.0000000000000343. PMID 24911353
- [Derived] Roy-Ghanta S, Van der Most R, Li P, Vaughn DW. Responses to A(H1N1)pdm09 influenza vaccines in participants previously vaccinated with seasonal influenza vaccine: a randomized, observer-blind, controlled study. J Infect Dis. 2014 Nov 1;210(9):1419-30. doi: 10.1093/infdis/jiu284. Epub 2014 May 26. PMID 24864125

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- GSK692342 Group: Subjects received 2 doses of the GSK692342 vaccine, intramuscularly into the deltoid region of the non-dominant arm, at Day 0 and into the deltoid region of the dominant arm, at Day 30.
- Control Group: Subjects received 2 doses of the GSK AS01E adjuvant, intramuscularly into the deltoid region of the non-dominant arm, at Day 0 and into the deltoid region of the dominant arm, at Day 30.
- Placebo Group: Subjects received 2 doses of saline solution, intramuscularly into the deltoid region of the non-dominant arm, at Day 0 and into the deltoid region of the dominant arm, at Day 30.
Period: Overall Study
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Started | 22 | 8 | 7
Completed | 22 | 8 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK692342 Group | Control Group | Placebo Group | Total
Number analyzed (Participants) | 22 | 8 | 7 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.6 (7.43) | 40.0 (5.61) | 41.9 (4.67) | 40.12 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 0 | 11
  Male | 14 | 5 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: During the 7-day period (Days 0-6) post vaccination following each dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  Any Pain, Dose 1 | 20 | 6 | 1
  Grade 3 Pain, Dose 1 | 1 | 0 | 0
  Any Redness, Dose 1 | 9 | 2 | 0
  Grade 3 Redness, Dose 1 | 2 | 0 | 0
  Any Swelling, Dose 1 | 8 | 1 | 0
  Grade 3 Swelling, Dose 1 | 2 | 0 | 0
  Any Pain, Dose 2 | 20 | 7 | 2
  Grade 3 Pain, Dose 2 | 3 | 0 | 0
  Any Redness, Dose 2 | 8 | 0 | 0
  Grade 3 Redness, Dose 2 | 0 | 0 | 0
  Any Swelling, Dose 2 | 7 | 1 | 0
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0
  Any Pain, Across | 21 | 8 | 3
  Grade 3 Pain, Across | 4 | 0 | 0
  Any Redness, Across | 13 | 2 | 0
  Grade 3 Redness, Across | 2 | 0 | 0
  Any Swelling, Across | 10 | 2 | 0
  Grade 3 Swelling, Across | 2 | 0 | 0

2. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastrointestinal symptoms (gastro) [nausea, vomiting, diarrhoea and/or abdominal pain], headache, malaise and myalgia. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day period (Days 0-6) post vaccination following each dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  Any Fatigue, Dose 1 | 10 | 6 | 2
  Grade 3 Fatigue, Dose 1 | 1 | 0 | 0
  Related Fatigue, Dose 1 | 0 | 0 | 0
  Any Gastro, Dose 1 | 4 | 2 | 1
  Grade 3 Gastro, Dose 1 | 0 | 0 | 0
  Related Gastro, Dose 1 | 0 | 0 | 0
  Any Headache, Dose 1 | 7 | 4 | 2
  Grade 3 Headache, Dose 1 | 0 | 0 | 0
  Related Headache, Dose 1 | 0 | 0 | 0
  Any Malaise, Dose 1 | 3 | 1 | 0
  Grade 3 Malaise, Dose 1 | 1 | 0 | 0
  Related Malaise, Dose 1 | 0 | 0 | 0
  Any Myalgia, Dose 1 | 3 | 2 | 0
  Grade 3 Myalgia, Dose 1 | 0 | 0 | 0
  Related Myalgia, Dose 1 | 0 | 0 | 0
  Any Temperature, Dose 1 | 0 | 1 | 1
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0
  Related Temperature, Dose 1 | 0 | 0 | 0
  Any Fatigue, Dose 2 | 18 | 3 | 2
  Grade 3 Fatigue, Dose 2 | 1 | 0 | 0
  Related Fatigue, Dose 2 | 0 | 0 | 0
  Any Gastro, Dose 2 | 4 | 2 | 0
  Grade 3 Gastro, Dose 2 | 1 | 0 | 0
  Related Gastro, Dose 2 | 0 | 0 | 0
  Any Headache, Dose 2 | 11 | 3 | 2
  Grade 3 Headache, Dose 2 | 1 | 0 | 0
  Related Headache, Dose 2 | 0 | 0 | 0
  Any Malaise, Dose 2 | 3 | 1 | 1
  Grade 3 Malaise, Dose 2 | 0 | 0 | 0
  Related Malaise, Dose 2 | 0 | 0 | 0
  Any Myalgia, Dose 2 | 6 | 1 | 1
  Grade 3 Myalgia, Dose 2 | 0 | 0 | 1
  Related Myalgia, Dose 2 | 0 | 0 | 0
  Any Temperature, Dose 2 | 5 | 1 | 0
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0
  Related Temperature, Dose 2 | 0 | 0 | 0
  Any Fatigue, Across | 18 | 6 | 3
  Grade 3 Fatigue, Across | 1 | 0 | 0
  Related Fatigue, Across | 0 | 0 | 0
  Any Gastro, Across | 7 | 3 | 1
  Grade 3 Gastro, Across | 1 | 0 | 0
  Related Gastro, Across | 0 | 0 | 0
  Any Headache, Across | 13 | 4 | 3
  Grade 3 Headache, Across | 1 | 0 | 0
  Related Headache, Across | 0 | 0 | 0
  Any Malaise, Across | 6 | 1 | 1
  Grade 3 Malaise, Across | 1 | 0 | 0
  Related Malaise, Across | 0 | 0 | 0
  Any Myalgia, Across | 7 | 2 | 1
  Grade 3 Myalgia, Across | 0 | 0 | 1
  Related Myalgia, Across | 0 | 0 | 0
  Any Temperature, Across | 5 | 2 | 1
  Grade 3 Temperature, Across | 0 | 0 | 0
  Related Temperature, Across | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day period (Days 0-29) post vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  Any AEs | 21 | 6 | 5
  Grade 3 AEs | 11 | 2 | 0
  Related AEs | 4 | 0 | 0

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity
Time Frame: During the entire study period, from Day 0 up to Day 210
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects | 2 | 0 | 0

5. Primary Outcome: Number of Subjects With Normal Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALT], aspartate aminotransferase [AST], basophils [BAS], creatinine [CREA], eosinophil [EOS]. Levels of haematological/biochemical parameters assessed in relation to normal laboratory values were - normal, below and above.
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  ALT, Day 0-normal | 17 | 5 | 7
  ALT, Day 7-normal | 16 | 4 | 7
  ALT, Day 30-normal | 16 | 5 | 7
  ALT, Day 37-normal | 16 | 6 | 6
  ALT, Day 60-normal | 15 | 7 | 7
  AST, Day 0-normal | 13 | 6 | 7
  AST, Day 7-normal | 11 | 6 | 4
  AST, Day 30-normal | 11 | 4 | 5
  AST, Day 37-normal | 12 | 5 | 5
  AST, Day 60-normal | 13 | 6 | 6
  BAS, Day 0-normal | 19 | 8 | 5
  BAS, Day 7-normal | 20 | 8 | 6
  BAS, Day 30-normal | 18 | 8 | 5
  BAS, Day 37-normal | 12 | 8 | 7
  BAS, Day 60-normal | 18 | 7 | 5
  CREA, Day 0-normal | 21 | 7 | 6
  CREA, Day 7-normal | 20 | 8 | 7
  CREA, Day 30-normal | 20 | 7 | 6
  CREA, Day 37-normal | 19 | 7 | 6
  CREA, Day 60-normal | 21 | 7 | 6
  EOS, Day 0-normal | 16 | 7 | 6
  EOS, Day 7-normal | 18 | 7 | 7
  EOS, Day 30-normal | 20 | 7 | 4
  EOS, Day 37-normal | 17 | 7 | 5
  EOS, Day 60-normal | 16 | 6 | 7

6. Primary Outcome: Number of Subjects With Normal Haematological Levels
Description: Among biochemical and haematological parameters assessed were haematocrit [Hct], haemoglobin [Hgb], lymphocytes [LYM], monocytes [MON], neutrophils [NEU]. Levels of haematological/biochemical parameters assessed in relation to normal laboratory values were - normal, below and above.
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  Hct, Day 0-normal | 18 | 6 | 7
  Hct, Day 7-normal | 18 | 6 | 7
  Hct, Day 30-normal | 20 | 8 | 7
  Hct, Day 37-normal | 16 | 6 | 7
  Hct, Day 60-normal | 18 | 8 | 7
  Hgb, Day 0-normal | 19 | 8 | 7
  Hgb, Day 7-normal | 15 | 7 | 7
  Hgb, Day 30-normal | 18 | 8 | 7
  Hgb, Day 37-normal | 18 | 7 | 7
  Hgb, Day 60-normal | 17 | 8 | 7
  LYM, Day 0-normal | 12 | 6 | 7
  LYM, Day 7-normal | 16 | 6 | 7
  LYM, Day 30-normal | 12 | 6 | 6
  LYM, Day 37-normal | 18 | 6 | 6
  LYM, Day 60-normal | 16 | 6 | 7
  MON, Day 0-normal | 21 | 8 | 6
  MON, Day 7-normal | 21 | 8 | 6
  MON, Day 30-normal | 21 | 8 | 7
  MON, Day 37-normal | 21 | 8 | 6
  MON, Day 60-normal | 22 | 7 | 6
  NEU, Day 0-normal | 14 | 7 | 5
  NEU, Day 7-normal | 21 | 7 | 7
  NEU, Day 30-normal | 17 | 7 | 7
  NEU, Day 37-normal | 16 | 7 | 6
  NEU, Day 60-normal | 16 | 7 | 7

7. Primary Outcome: Number of Subjects With Normal Haematological Levels
Description: Among biochemical and haematological parameters assessed were platelets [PLA], red blood cells [RBC] and white blood cells [WBC]. Levels of haematological/biochemical parameters assessed in relation to normal laboratory values were - normal, below and above.
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  PLA, Day 0-normal | 21 | 7 | 5
  PLA, Day 7-normal | 21 | 8 | 5
  PLA, Day 30-normal | 21 | 6 | 4
  PLA, Day 37-normal | 21 | 7 | 5
  PLA, Day 60-normal | 20 | 7 | 4
  RBC, Day 0-normal | 13 | 5 | 6
  RBC, Day 7-normal | 13 | 5 | 6
  RBC, Day 30-normal | 13 | 6 | 6
  RBC, Day 37-normal | 12 | 6 | 5
  RBC, Day 60-normal | 13 | 7 | 6
  WBC, Day 0-normal | 16 | 7 | 5
  WBC, Day 7-normal | 18 | 7 | 5
  WBC, Day 30-normal | 16 | 6 | 6
  WBC, Day 37-normal | 17 | 6 | 5
  WBC, Day 60-normal | 16 | 6 | 5

8. Primary Outcome: Number of Subjects With Biochemical and Haematological Levels Below Normal
Description: as for outcome 5
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  ALT, Day 0-below | 1 | 0 | 0
  ALT, Day 7-below | 0 | 0 | 0
  ALT, Day 30-below | 1 | 0 | 0
  ALT, Day 37-below | 1 | 0 | 0
  ALT, Day 60-below | 1 | 0 | 0
  AST, Day 0-below | 0 | 0 | 0
  AST, Day 7-below | 0 | 0 | 0
  AST, Day 30-below | 0 | 0 | 0
  AST, Day 37-below | 0 | 0 | 0
  AST, Day 60-below | 0 | 0 | 0
  BAS, Day 0-below | 1 | 0 | 1
  BAS, Day 7-below | 0 | 0 | 1
  BAS, Day 30-below | 2 | 0 | 0
  BAS, Day 37-below | 5 | 0 | 0
  BAS, Day 60-below | 1 | 1 | 2
  CREA, Day 0-below | 0 | 1 | 1
  CREA, Day 7-below | 0 | 0 | 0
  CREA, Day 30-below | 1 | 1 | 1
  CREA, Day 37-below | 0 | 1 | 0
  CREA, Day 60-below | 0 | 1 | 1
  EOS, Day 0-below | 4 | 1 | 1
  EOS, Day 7-below | 3 | 1 | 0
  EOS, Day 30-below | 0 | 1 | 3
  EOS, Day 37-below | 4 | 1 | 1
  EOS, Day 60-below | 4 | 1 | 0

9. Primary Outcome: Number of Subjects With Haematological Levels Below Normal
Description: as for outcome 6
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  Hct, Day 0-below | 4 | 2 | 0
  Hct, Day 7-below | 4 | 2 | 0
  Hct, Day 30-below | 2 | 0 | 0
  Hct, Day 37-below | 6 | 2 | 0
  Hct, Day 60-below | 4 | 0 | 0
  Hgb, Day 0-below | 3 | 0 | 0
  Hgb, Day 7-below | 7 | 1 | 0
  Hgb, Day 30-below | 4 | 0 | 0
  Hgb, Day 37-below | 4 | 1 | 0
  Hgb, Day 60-below | 5 | 0 | 0
  LYM, Day 0-below | 10 | 2 | 0
  LYM, Day 7-below | 6 | 2 | 0
  LYM, Day 30-below | 10 | 2 | 0
  LYM, Day 37-below | 4 | 2 | 0
  LYM, Day 60-below | 6 | 2 | 0
  MON, Day 0-below | 1 | 0 | 0
  MON, Day 7-below | 1 | 0 | 0
  MON, Day 30-below | 1 | 0 | 0
  MON, Day 37-below | 1 | 0 | 0
  MON, Day 60-below | 0 | 0 | 0
  NEU, Day 0-below | 7 | 1 | 0
  NEU, Day 7-below | 1 | 1 | 0
  NEU, Day 30-below | 5 | 1 | 0
  NEU, Day 37-below | 5 | 1 | 0
  NEU, Day 60-below | 5 | 1 | 0

10. Primary Outcome: Number of Subjects With Haematological Levels Below Normal
Description: Among biochemical and haematological parameters assessed were [PLA], red blood cells [RBC] and white blood cells [WBC]. Levels of haematological/biochemical parameters assessed in relation to normal laboratory values were - normal, below and above.
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  PLA, Day 0-below | 1 | 1 | 1
  PLA, Day 7-below | 1 | 0 | 1
  PLA, Day 30-below | 1 | 1 | 2
  PLA, Day 37-below | 1 | 1 | 1
  PLA, Day 60-below | 1 | 1 | 2
  RBC, Day 0-below | 9 | 3 | 1
  RBC, Day 7-below | 9 | 3 | 1
  RBC, Day 30-below | 9 | 2 | 1
  RBC, Day 37-below | 10 | 2 | 2
  RBC, Day 60-below | 9 | 1 | 1
  WBC, Day 0-below | 5 | 1 | 0
  WBC, Day 7-below | 4 | 1 | 0
  WBC, Day 30-below | 6 | 2 | 0
  WBC, Day 37-below | 4 | 1 | 0
  WBC, Day 60-below | 5 | 2 | 0

11. Primary Outcome: Number of Subjects With Biochemical and Haematological Levels Above Normal
Description: as for outcome 5
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  ALT, Day 0-above | 4 | 3 | 0
  ALT, Day 7-above | 6 | 4 | 0
  ALT, Day 30-above | 5 | 3 | 0
  ALT, Day 37-above | 5 | 2 | 1
  ALT, Day 60-above | 6 | 1 | 0
  AST, Day 0-above | 9 | 2 | 0
  AST, Day 7-above | 11 | 2 | 3
  AST, Day 30-above | 11 | 4 | 2
  AST, Day 37-above | 10 | 3 | 2
  AST, Day 60-above | 9 | 2 | 1
  BAS, Day 0-above | 2 | 0 | 1
  BAS, Day 7-above | 2 | 0 | 0
  BAS, Day 30-above | 2 | 0 | 2
  BAS, Day 37-above | 5 | 0 | 0
  BAS, Day 60-above | 3 | 0 | 0
  CREA, Day 0-above | 1 | 0 | 0
  CREA, Day 7-above | 2 | 0 | 0
  CREA, Day 30-above | 1 | 0 | 0
  CREA, Day 37-above | 3 | 0 | 1
  CREA, Day 60-above | 1 | 0 | 0
  EOS, Day 0-above | 2 | 0 | 0
  EOS, Day 7-above | 1 | 0 | 0
  EOS, Day 30-above | 2 | 0 | 0
  EOS, Day 37-above | 1 | 0 | 1
  EOS, Day 60-above | 2 | 1 | 0

12. Primary Outcome: Number of Subjects With Haematological Levels Above Normal
Description: as for outcome 6
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  Hct, Day 0-above | 0 | 0 | 0
  Hct, Day 7-above | 0 | 0 | 0
  Hct, Day 30-above | 0 | 0 | 0
  Hct, Day 37-above | 0 | 0 | 0
  Hct, Day 60-above | 0 | 0 | 0
  Hgb, Day 0-above | 0 | 0 | 0
  Hgb, Day 7-above | 0 | 0 | 0
  Hgb, Day 30-above | 0 | 0 | 0
  Hgb, Day 37-above | 0 | 0 | 0
  Hgb, Day 60-above | 0 | 0 | 0
  LYM, Day 0-above | 0 | 0 | 0
  LYM, Day 7-above | 0 | 0 | 0
  LYM, Day 30-above | 0 | 0 | 1
  LYM, Day 37-above | 0 | 0 | 1
  LYM, Day 60-above | 0 | 0 | 0
  MON, Day 0-above | 0 | 0 | 1
  MON, Day 7-above | 0 | 0 | 1
  MON, Day 30-above | 0 | 0 | 0
  MON, Day 37-above | 0 | 0 | 1
  MON, Day 60-above | 0 | 1 | 1
  NEU, Day 0-above | 1 | 0 | 2
  NEU, Day 7-above | 0 | 0 | 0
  NEU, Day 30-above | 0 | 0 | 0
  NEU, Day 37-above | 1 | 0 | 1
  NEU, Day 60-above | 1 | 0 | 0

13. Primary Outcome: Number of Subjects With Haematological Levels Above Normal
Description: as for outcome 10
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects
  PLA, Day 0-above | 0 | 0 | 1
  PLA, Day 7-above | 0 | 0 | 1
  PLA, Day 30-above | 0 | 1 | 1
  PLA, Day 37-above | 0 | 0 | 1
  PLA, Day 60-above | 1 | 0 | 1
  RBC, Day 0-above | 0 | 0 | 0
  RBC, Day 7-above | 0 | 0 | 0
  RBC, Day 30-above | 0 | 0 | 0
  RBC, Day 37-above | 0 | 0 | 0
  RBC, Day 60-above | 0 | 0 | 0
  WBC, Day 0-above | 1 | 0 | 2
  WBC, Day 7-above | 0 | 0 | 2
  WBC, Day 30-above | 0 | 0 | 1
  WBC, Day 37-above | 1 | 1 | 2
  WBC, Day 60-above | 1 | 0 | 2

14. Secondary Outcome: Frequency of Mycobacterium Tuberculosis Fusion Protein (M72) Specific Cluster of Differentiation 4/8 (CD4/8+) T Cells Expressing at Least Two Different Cytokines
Description: Among cytokines expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS).
Time Frame: At Day 0, 30, 60 and 210
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
T cells/million cells
  CD4-All Doubles, Day 0 [N=22;8;7] | 95.0 [1.0 to 218.0] | 154.5 [40.5 to 160.5] | 96.0 [1.0 to 267.0]
  CD4-All Doubles, Day 30 [N=22;8;7] | 1713.5 [507.0 to 2786.0] | 129.0 [103.5 to 204.5] | 94.0 [1.0 to 226.0]
  CD4-All Doubles, Day 60 [N=22;8;7] | 7003.5 [3691.0 to 10701.0] | 112.0 [51.0 to 258.0] | 26.0 [13.0 to 227.0]
  CD4-All Doubles, Day 210 [N=21;8;7] | 4245.0 [2427.0 to 6121.0] | 83.5 [16.0 to 140.0] | 67.0 [4.0 to 133.0]
  CD8-All Doubles, Day 0 [N=22;8;7] | 167.0 [1.0 to 358.0] | 71.5 [11.0 to 442.0] | 364.0 [80.0 to 1001.0]
  CD8-All Doubles, Day 30 [N=22;8;7] | 97.0 [27.0 to 507.0] | 38.5 [8.0 to 293.0] | 216.0 [1.0 to 986.0]
  CD8-All Doubles, Day 60 [N=22;8;7] | 236.0 [19.0 to 542.0] | 74.5 [1.0 to 570.0] | 415.0 [25.0 to 889.0]
  CD8-All Doubles, Day 210 [N=21;8;7] | 195.0 [20.0 to 340.0] | 55.5 [1.0 to 248.5] | 241.0 [39.0 to 858.0]

15. Secondary Outcome: Frequency of M72 Specific CD4/8+ T Cells Expressing at Least One Cytokine and Another Signal Molecule
Description: Expressed cytokine combinations for CD4+ T cells were CD40-L and interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α]; IL-2 and CD40-L, or IFN-γ, or TNF-α; IFN-γ and CD40-L, or IL-2, or TNF-α; TNF-α and CD40-L, or IL-2, or IFN-γ.
  For CD8+ T cells no vaccine induced responses were observed, thus results are presented only for the frequency of M72-specific CD8+ T cells expressing at least two cytokines.
Time Frame: At Day 0, 30, 60 and 210
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
T cells/million cells
  CD4-CD40-L, Day 0 [N=22;8;7] | 88.5 [26.0 to 185.0] | 135.0 [54.0 to 152.0] | 110.0 [1.0 to 240.0]
  CD4-CD40-L, Day 30 [N=22;8;7] | 1389.5 [506.0 to 2359.0] | 129.0 [71.5 to 196.5] | 94.0 [1.0 to 226.0]
  CD4-CD40-L, Day 60 [N=22;8;7] | 6771.5 [3334.0 to 10235.0] | 112.0 [54.5 to 211.5] | 40.0 [26.0 to 213.0]
  CD4-CD40-L, Day 210 [N=21;8;7] | 3953.0 [1477.0 to 4853.0] | 71.0 [1.0 to 145.0] | 53.0 [1.0 to 120.0]
  CD4-IL-2, Day 0 [N=22;8;7] | 104.0 [40.0 to 160.0] | 87.0 [52.5 to 118.0] | 120.0 [13.0 to 267.0]
  CD4-IL-2, Day 30 [N=22;8;7] | 1140.0 [427.0 to 2141.0] | 136.5 [58.0 to 200.0] | 93.0 [12.0 to 173.0]
  CD4-IL-2, Day 60 [N=22;9;7] | 6640.5 [3213.0 to 9520.0] | 80.0 [22.0 to 253.5] | 27.0 [1.0 to 174.0]
  CD4-IL-2, Day 210 [N=21;8;7] | 4166.0 [1477.0 to 5347.0] | 74.0 [1.0 to 127.0] | 67.0 [1.0 to 120.0]
  CD40-TNF-α, Day 0 [N=22;8;7] | 40.0 [1.0 to 120.0] | 106.5 [63.5 to 154.5] | 63.0 [1.0 to 240.0]
  CD4-TNF-α, Day 30 [N=22;8;7] | 793.5 [226.0 to 2093.0] | 27.5 [20.0 to 65.0] | 107.0 [13.0 to 147.0]
  CD4-TNF-α, Day 60 [N=22;8;7] | 4286.5 [2294.0 to 6880.0] | 38.5 [11.5 to 78.5] | 80.0 [13.0 to 226.0]
  CD4-TNF-α, Day 210 [N=21;8;7] | 2632.0 [1560.0 to 4186.0] | 54.0 [17.5 to 81.0] | 54.0 [13.0 to 107.0]
  CD40-IFN-γ, Day 0 [N=22;8;7] | 64.0 [26.0 to 212.0] | 29.5 [19.0 to 113.5] | 67.0 [26.0 to 147.0]
  CD4-IFN-γ, Day 30 [N=22;8;7] | 413.5 [119.0 to 1373.0] | 99.0 [82.5 to 147.5] | 106.0 [26.0 to 199.0]
  CD4-IFN-γ, Day 60 [N=22;8;7] | 1733.5 [440.0 to 3455.0] | 102.5 [53.0 to 221.0] | 26.0 [13.0 to 79.0]
  CD4-IFN-γ, Day 210 [N=21;8;7] | 667.0 [227.0 to 2026.0] | 51.5 [1.0 to 87.0] | 40.0 [1.0 to 119.0]

16. Secondary Outcome: Cell Count of CD4+ T Cells
Description: CD4+ T cell counts are defined by values greater than (>) 200 cells per cubic millimeters (mm3) at screening for enrolment into the study.
Time Frame: At Day 0, 30, 60 and 210
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: T cells/cubic millimeter
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
T cells/cubic millimeter
  CD4+ T Cells, Day 0 | 585 [416 to 651] | 437 [318.5 to 561] | 811 [704 to 1050]
  CD4+ T Cells, Day 30 | 566 [465 to 713] | 410.5 [283.5 to 527.5] | 799 [750 to 978]
  CD4+ T Cells, Day 60 | 567 [457 to 679] | 368 [339 to 572.5] | 877 [745 to 1062]
  CD 4+ T Cells, Day 210 | 548.5 [426 to 680] | 433 [377 to 534] | 822 [741 to 1138]

17. Secondary Outcome: Anti-M72 Specific Antibody Concentrations
Description: Concentrations given in Enzyme-Linked Immunosorbent Assay units per milliliter (EL.U/mL) were expressed in Geometric Mean Concentrations (GMCs).
Time Frame: At Day 0, 30, 60 and 210
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
EL.U/mL
  Anti-M72, Day 0 [N=22;8;7] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4]
  Anti-M72, Day 30 [N=22;8;7] | 2.1 [1.5 to 2.9] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4]
  Anti-M72, Day 60 [N=22;8;7] | 282.4 [177.2 to 450.0] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4]
  Anti-M72, Day 210 [N=21;8;7] | 38.3 [22.8 to 64.2] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4]

18. Secondary Outcome: Number of Subjects With Significant Highly Active Anti-Retroviral Therapy (HAART) Changes
Description: Recorded significant HAART change refers to one subject switching the Combivir drug to Truvada as planned by personal physician, with no relationship to vaccination, prior to study enrolment.
Time Frame: From Day 60 to Day 210
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Number analyzed (Participants) | 22 | 8 | 7
Subjects | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day period; Unsolicited AEs: during the 30-day period; SAEs: during the entire study period, from Day 0 up to Day 210.
Arm/Group | GSK692342 Group | Control Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 2/22 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 21/22 | 8/8 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK692342 Group (N=22) | Control Group (N=8) | Placebo Group (N=7)
Appendicitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK692342 Group (N=22) | Control Group (N=8) | Placebo Group (N=7)
Nasopharyngitis (Infections and infestations) | 4 | 2 | 2
Headache (Nervous system disorders) | 5 | 2 | 0
Cd4 lymphocytes decreased (Investigations) | 5 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Migraine (Nervous system disorders) | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Fatigue (General disorders) | 2 | 0 | 0
Feeling hot (General disorders) | 2 | 0 | 0
Injection site pruritus (General disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Pterygium (Eye disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pain (General disorders) | 21 | 8 | 3
Redness (General disorders) | 13 | 2 | 0
Swelling (General disorders) | 10 | 2 | 0
Fatigue (General disorders) | 18 | 6 | 3 — Solicited general symptom
Gastrointestinal (General disorders) | 7 | 3 | 1
Headache (General disorders) | 13 | 4 | 3 — Solicited general symptom
Malaise (General disorders) | 6 | 1 | 1
Myalgia (General disorders) | 7 | 2 | 1
Temperature (Axillary) (General disorders) | 5 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.